CLINICAL TRIAL: NCT06394661
Title: Serplulimab Combined With NabPE for Early-stage Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative (HR+/HER2-) Breast Cancer- A Single-arm, Multicenter, Phase 2 Clinical Study
Brief Title: Serplulimab Plus Chemotherapy for Early-stage HR+/HER2- Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-018
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: HR+ breast cancer; neoadjuvant; serplulimab
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Serplulimab group (Experimental): NabPE+Serplulimab group（Epirubicin 75mg/m2 ivgtt on Day 1+Albumin Paclitaxel 260mg/m2 ivgtt on Day 1+Serplulimab 4.5mg/Kg ivgtt on Day 3）every 3 weeks for 6 cycles. Then paticipants will receive surgery and Serplulimab will be given as monotherapy every 3 weeks up to 6 months from the beginning of the treatment.
  Interventions: Drug: Serplulimab+NabPE

INTERVENTIONS:
Drug: Serplulimab+NabPE — Serplulimab plus neoadjuvant nab-PE: Epirubicin 75mg/m2 ivgtt on Day 1+Albumin Paclitaxel 260mg/m2 ivgtt on Day 1+Serplulimab 4.5mg/Kg ivgtt on Day 3）

SUMMARY:
The goal of this clinical trial is to learn if serplulimab is effective in early HR+/HER2- breast cancer. It will also learn about the safety of serplulimab. The main questions it aims to answer are:

Does serplulimab combined with neoadjuvant chemotherapy improve the pCR rate of early HR+/HER2- breast cancer? What medical problems do participants have when receiving serplulimab? Researchers will compare the effect of serplulimab combined with chemotherapy to the effect of chemotherapy reported in literature.

Participants will: Receive serplulimab plus chemotherapy every 3 weeks for 6 cycles; All patients will receive surgery, and the primary end point is a pathological complete response at the time of definitive surgery; After definitive surgery, the participants will receive adjuvant serplulimab every 3 weeks for up to 6 months from the beginning of the treatment.

DETAILED DESCRIPTION:
In recent years, significant progress has been made in the immunotherapy of breast cancer, and PD1/PDL1 inhibitors have achieved good results in the treatment of triple-negative breast cancer. There have also been many attempts to apply them in HR+/HER2- breast cancer. In the I-SPY2 study, Pembrolizumab combined with chemotherapy increased the pCR rate of HR+/HER2- breast cancer from 13% in the chemotherapy alone group to 30%. In the KEYNOTE756 study, Pembrolizumab in combination with chemotherapy increased the pCR rate by 8.5% (24.3% vs. 15.6%) compared to the chemotherapy-only arm in HR+/HER2- breast cancer. pCR rates in the Nivolumab arm of the CheckMate 7FL study were 24.5% compared with 13.8% in the control arm. While further long-term follow-up data are still needed to confirm patient benefit, it still provides a new treatment option for HR+/HER2- breast cancer patients.

The neoadjuvant treatment options commonly used for HR+/HER2- breast cancer are mainly anthracycline sequential or combined with paclitaxel chemotherapy regimens. Several clinical studies have confirmed that albumin paclitaxel is more effective than solvent-based paclitaxel, and therefore, albumin paclitaxel in combination with epirubicin has also become a commonly used chemotherapy regimen in clinical practice.

The aim of this study was to explore the efficacy and safety of the Serplulimab combined with nab-paclitaxel and epirubicin in the neoadjuvant treatment of HR+/HER2- breast cancer

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following criteria to be eligible:

Age: ≥18 years old.

Clinical-pathological confirmation:

cT2-cT4 breast cancer, or cT1c with axillary lymph node metastasis.

Histopathologically confirmed HR+/HER2- invasive breast cancer:

ER and/or PR positive (IHC nuclear staining ≥1%).

HER2-negative (IHC 0 or 1+ without FISH testing, or IHC 2+ with FISH-negative amplification).

Ki67 ≥20%.

Clinically measurable lesions:

Measurable lesions confirmed by ultrasound, mammography, or MRI (optional) within 1 month prior to randomization.

Adequate organ and bone marrow function (within 1 month prior to chemotherapy):

Absolute neutrophil count (ANC) ≥2.0 × 10^9/L.

Hemoglobin ≥90 g/L.

Platelet count ≥100 × 10^9/L.

Total bilirubin <1.5 × ULN (upper limit of normal).

Creatinine <1.5 × ULN.

AST/ALT <1.5 × ULN.

Cardiac function: Left ventricular ejection fraction (LVEF) ≥55% by echocardiography.

Reproductive status: Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomization.

ECOG performance status: ≤1.

Informed consent: Signed written informed consent.

Exclusion Criteria

Patients meeting any of the following criteria will be excluded:

Evidence of metastatic breast cancer:

Prior systemic therapy: Chemotherapy, endocrine therapy, targeted therapy, or radiotherapy for the current breast cancer.

Second primary malignancy, except: Adequately treated non-melanoma skin cancer.

Prior immunotherapy: Treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or other immune checkpoint inhibitors.

Immune-related conditions:

Diagnosed immunodeficiency or active autoimmune disease.

Severe cardiopulmonary disease: Uncontrolled or clinically significant.

Active hepatitis B or C.

Pregnancy or lactation: Pregnant or breastfeeding women.

Other contraindications: Severe uncontrolled comorbidities deemed by investigators to contraindicate chemotherapy or PD-1 inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2024-04-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | up to 24 weeks
  After neoadjuvant chemotherapy and surgery, the resected specimen (breast + axilla) was free of any invasive cancer (ie, ypT0/is, ypN0)

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5-10 years
  EFS was defined as the time from randomization to any of the following events: disease progression during neoadjuvant therapy, local or distant recurrence, second primary malignancy (breast or other cancer), or death from any cause.
DFS | 5-10 years
  Disease-free Survival,From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause
Objective Response Rate (ORR) | up to 24 weeks
  ORR is defined as proportion of patients demonstrating either a partial response (PR) or a complete response (CR)
adverse events | After each cycle of chemotherapy (21 days as 1 cycle)]
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

OTHER OUTCOMES:
PDL1 expression | up to 24 weeks
  Evaluate the impact of PDL1 expression on treatment efficacy
next-generation sequencing (NGS) | up to 24 weeks
  NGS analysis to identify genetic alterations that predict response to anti-PD1 treatment
blood based biomarker | up to 24 weeks
  To evaluate blood based biomarkers include immune cell subsets and cytokines.
9-item depression module of the Patient Health Questionnaire-9 | up to 24 weeks
  PHQ-9 questionnaire to evaluate level of depression of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, PhD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cacer hospital, Henan, Henan, China

IPD SHARING:
Plan to Share IPD: No